CLINICAL TRIAL: NCT04289272
Title: A Pilot Randomised Control Trial to Examine the Acceptability, Feasibility, and Efficacy of 'Confident Me' School Workshops for Body Confidence in India
Brief Title: Evaluating Dove Confident Me in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Lady Shri Ram College for Women (Unknown); Tata Institute of Social Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAS.18.01.074
Record Dates: First submitted 2020-02-05; First posted 2020-02-28 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Body Image
Keywords: body image; school; intervention; adolescence; self-esteem

STUDY DESIGN:
Intervention Model Description: Parallel 2-arm cluster randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: masking not possible for participants within design, but outcome assessors do not know which condition participants are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dove Confident Me (Experimental): Dove Confident Me body image intervention to be delivered to students 1 lesson per week for 5 weeks (5 x 45 minute lessons).
  Interventions: Behavioral: Dove Confident Me
- Control (No Intervention): Students receive lessons-as-usual.

INTERVENTIONS:
Behavioral: Dove Confident Me — Dove Confident Me is a school-based intervention co-created by researchers at La Trobe University (Australia), the Centre for Appearance Research UWE, teachers, students, and education experts, and the Dove Self-Esteem Project (the social mission for personal care brand Dove). The five-session intervention is aimed at adolescents aged between 11-13 years, and targets recognised risk factors for body dissatisfaction, by addressing societal appearance ideals (Session 1), media literacy (Session 2), appearance comparisons (Session 3), appearance-related conversations and teasing (Session 4), and promoting 'body activism' (Session 5). The intervention consists of classroom-based discussion and small group activities, and uses audio-visual materials and worksheets to facilitate learning.
  Arms: Dove Confident Me

SUMMARY:
Body image is one of the leading concerns for young people. Such concerns can have serious health consequences, including unhealthy weight control and exercise behaviours, depression and self-harm, low self-esteem and substance abuse. Emerging approaches for improving body image are effective among adolescent girls and boys in the school setting. However, the vast majority of trials in this area are conducted in high-income westernised countries, despite body image concerns increasingly being recognised as a global concern. As such, it is important to develop and disseminate interventions to promote positive body image among adolescents in in low-to-middle income countries, too. 'Confident Me' has been found to be effective in improving body image and related outcomes among adolescent girls and boys in the UK up to 12-months later, and thus, could undergo adaptations for the Indian context.

The aim of the present study is two-fold:

* To conduct a small-scale acceptability study of a 'Confident Me', a body image intervention, among 11-13-year olds in New Delhi, India, to understand its acceptability, feasibility, and preliminary efficacy in a metropolitan area of India.
* To refine 'Confident Me' based on the acceptability study, and to conduct a randomised controlled trial to evaluate its efficacy at improving body image and related outcomes among 11-13-year olds in New Delhi, India.

The first aim will be fulfilled by recruiting two schools, of which one will be randomised to the intervention and the other to the control arm. We will compare the body image and well-being of students who take part in the programme to students in the control group. The investigators will also gather in-depth feedback from students, teachers and the interventionist via focus groups and interviews, in order to inform future improvement of the programme. The second aim will be fulfilled by randomising six schools to either the revised body image programme (3 schools) or the control arm (3 schools). Students will complete questionnaire assessments of body image and well-being before and after the 5-week programme period, and again 12 weeks later to assess longer-term benefits.

DETAILED DESCRIPTION:
Background:

Body image is a significant and prevalent concern for adolescents in high-income countries such as the UK, the USA, and Australia. For example, a study of 1,600 girls in the UK found that four in ten 11-16-year-old girls are unhappy with the way they look. Similarly, a nationally representative survey of nearly 22,000 young people in Australia found that 3 in 10 adolescent boys and girls are very concerned about their body image, and body image was voted among the top three life concerns. The high prevalence of body image concerns among adolescent boys and girls is worrisome, given their serious negative physical and psychological health consequences. For example, body dissatisfaction is associated with engagement in unhealthy weight loss behaviours and the onset of eating disorders, depression and self-harm, substance use, and lower levels of academic engagement.

There is increasing recognition that body image is a global issue, as opposed to one relegated to privileged adolescents in high-income Westernised countries. For example, in India, 57% of adolescents aged 15-19 years report being concerned with their appearance. Further, adolescent girls across different regions of India have expressed concerns in relation to their weight and report dieting behaviours. Skin colour has also been indicated as an additional source of appearance concern among young people in India. A large-scale study among Asian, African, and South American countries, found that 19% of Indian undergraduate students had used a skin lightening product in the previous 12 months, strongly suggesting dissatisfaction with their natural skin tone, which may be pertinent to younger groups.

Collectively, these findings indicate the importance of developing and disseminating interventions to promote positive body image among adolescents in India. To date, only one published study has investigated the effectiveness of a body image intervention delivered in schools to adolescents in India. The results indicated the potential for media literacy to improve body satisfaction among adolescent girls. While this study offers a promising first step, more research is needed to understand the potential for school body image interventions in India.

The aim of the present study is two-fold:

1. To conduct a small-scale acceptability study of a body image intervention among 11-13-year olds in New Delhi, India, to understand its acceptability, feasibility, and preliminary efficacy in a metropolitan area of India.
2. To refine the body image intervention based on the acceptability study, and to conduct a randomised controlled trial to evaluate its efficacy at improving body image and related outcomes among 11-13-year olds in New Delhi, India.

1) The Acceptability Study

Design:

Two schools will be randomly allocated to receive the body image intervention or classes-as-usual (control). Students will be assessed on body image and related outcomes at baseline, post-intervention and 10 weeks follow-up, under standardised conditions.

Participants & recruitment:

Two co-educational secondary schools in Delhi, India, will be invited to take part in this study. The collaborators in India will recruit the schools, and they will likely be schools with which their institution has existing relations with. All students in classes 6-7 (equivalent of UK years 7-8; students aged 11-13) in each school will be invited to take part.

After expressing initial interest, each school will receive detailed information regarding the aims, objective and requirements of the study to help them decide if they would like to take part in this research project. In line with the ethical procedures adopted at the collaborators' Indian universities, the school's head teacher will provide active informed consent. Students will also be required to provide their consent before taking part. All students will have the opportunity to opt out of the study, or withdraw from the study at any time, irrespective of head teacher consent. The Indian ethical procedures do not involve asking parents to provide consent for their child's participation in the research.

The exact numbers of students that take part in this research will depend on the number of children enrolled in classes 6-7 at each school recruited, and the number that opt out during the student consent process or are lost at follow-up due to moving schools, or being away from school on the day the data is collected. However, given that this is a preliminary acceptability study, both conditions (i.e., schools) will include 80 girls and 80 boys (160 participants overall) aged 11 to 13 years, which allows for 30% attrition.

Intervention:

Dove Confident Me

Dove Confident Me is a school-based intervention co-created by researchers at La Trobe University (Australia), the Centre for Appearance Research UWE, teachers, students, and education experts, and the Dove Self-Esteem Project (the social mission for personal care brand Dove). The five-session intervention is aimed at adolescents aged between 11-13 years, and targets recognised risk factors for body dissatisfaction, by addressing societal appearance ideals (Session 1), media literacy (Session 2), appearance comparisons (Session 3), appearance-related conversations and teasing (Session 4), and promoting 'body activism' (Session 5). The intervention consists of classroom-based discussion and small group activities and uses audio-visual materials and worksheets to facilitate learning. The content is based upon an evidence-based intervention previously trialled among adolescent girls (Richardson and Paxton, 2010).

A large-scale cluster randomised controlled trial (RCT) evaluating Dove Confident Me found it to be effective in improving body image and related outcomes among adolescent girls and boys in the UK up to 12-months later when delivered by teachers (Diedrichs et al., under review). These findings present the longest improvements in body image observed in a teacher-led intervention. However, the intervention has not undergone evaluation in low- and middle- income countries, such as India, where body image concerns are also prevalent but the rigorous development, evaluation, and dissemination, of evidence-based interventions is lacking.

Procedure:

Investigators from the Centre for Appearance Research (CAR) based at the University of the West of England will be leading the study remotely from Bristol, UK. CAR researchers will be responsible for designing the study, analysing the data, and writing up the manuscript. They will also be working with Indian collaborators who will be responsible for translating the measures, recruiting the schools, collecting data, and delivering the intervention.

Students aged 11-13 from a further two secondary schools in Delhi will be recruited, and independent randomisation will be used to assign one school to the intervention condition, and the other to the lessons-as-usual control condition. This will be done using freely available computer software. Dove Confident Me (culturally adapted and translated into Hinglish) will be delivered by counselling psychologists at Karma Centre for Wellbeing in Delhi. The interventionists will be trained (in person) by two researchers from CAR on the delivery of the intervention. Both of these researchers possess experience of delivering, and training others to deliver, a range of body image interventions, including Dove Confident Me.

A questionnaire comprising the self-report measures described below will be used to assess the impact of the intervention on students' body image and associated risk factors. After obtaining consent from the school head teachers, and the students, these measures will be administered in the classroom to the 11-13 year old students at pre-intervention (1-2 weeks before intervention delivery), immediately after intervention delivery (within 1 week of the final session), and again at 10 weeks follow-up. The questionnaire will take students no more than 20-25 minutes to complete. Students will complete questionnaires under standardised conditions supervised by their teachers and trained research staff. Blinding of students, teachers, and researchers is not possible due to the nature of the intervention. However, risk of bias from teachers and researchers is minimised due to anonymous self-report assessments. Risk of contagion is also minimised by randomising at the school level. Participating schools will receive a £150 honorarium. This project has received ethical approval from the University of the West of England's Faculty Research Ethics Committee.

In order to assess the fidelity of the intervention manuals, all sessions will be audio-recorded as well as observed by a researcher and rated based on adherence to lesson plans. The interventionist and observing teachers also will be asked to complete a brief form after each lesson stating which activities were completed.

To assess intervention feasibility and acceptability, phone calls will be conducted with the interventionists after every session, to collect 'in-the-moment' feedback and suggestions for improvement to the materials. At the conclusion of the intervention, interviews will be conducted with the interventionists to explore their experience of delivering the body image lessons. They will also be asked how well the content of the intervention was received, how comfortable they felt delivering the session, and their suggestions to improve the intervention further. Class teachers observing the lessons will also be interviewed and asked similar questions.

In the post-intervention questionnaire, students will be asked a series of questions to assess their acceptability of the intervention. Students will indicate agreement with different statements using a 5-point Likert scale, and will be asked three open-ended questions: what they liked, what they did not like, and to list three things they learnt from the intervention. Additionally, a sub-sample of students (approximately 10 girls, 10 boys) in the intervention condition will also be invited to take part in single-gender focus groups, in order to explore their opinions of the intervention. Permission to audio record the focus groups and interviews will be sought from participants prior to commencing the discussions.

The findings from this study will then be used to refine the intervention material further, to ensure that it is adequately localised to the Indian context.

2) The Randomised Controlled Trial

Design:

Six schools will be randomly allocated to receive the body image intervention or classes-as-usual (control). Students will be assessed on body image and related outcomes at baseline, post-intervention and 12 weeks follow-up, under standardised conditions.

Participants & recruitment:

Six co-educational secondary schools in Delhi, India, will be invited to take part in this study. The collaborators in India will recruit the schools, and they will likely be schools with which their institution has existing relations with. All students in classes 6-8 (equivalent of UK years 7-9; students aged 11-14) in each school will be invited to take part.

After expressing initial interest, each school will receive detailed information regarding the aims, objective and requirements of the study to help them decide if they would like to take part in this research project. In line with the ethical procedures adopted at the collaborators' Indian universities, the school's head teacher will provide active informed consent. Students will also be required to provide their consent before taking part. All students will have the opportunity to opt out of the study, or withdraw from the study at any time, irrespective of head teacher consent. The Indian ethical procedures do not involve asking parents to provide consent for their child's participation in the research.

The exact numbers of students that take part in this research will depend on the number of children enrolled in classes 6-8 at each school recruited, and the number that opt out during the student consent process or are lost at follow-up due to moving schools, or being away from school on the day the data is collected. However, we will endeavour to include 125 girls and 125 boys (250 participants overall) aged 11 to 14 years, which allows for 30% attrition.

Procedure:

Students aged 11-14 from a further six secondary schools in Delhi will be recruited, and independent randomisation will be used to assign three schools to the intervention condition, and the other three to the lessons-as-usual control condition. This will be done using freely available computer software. The refined programme will be delivered by counselling psychologists at Karma Centre for Wellbeing in Delhi. The interventionists will be trained (in person) by two researchers from CAR on the delivery of the intervention. Both of these researchers possess experience of delivering, and training others to deliver, a range of body image interventions, including Dove Confident Me.

A questionnaire comprising the self-report measures described below will be used to assess the impact of the intervention on students' body image and associated risk factors. After obtaining consent from the school head teachers, and the students, these measures will be administered in the classroom to the 11-14 year old students at pre-intervention (1-2 weeks before intervention delivery), immediately after intervention delivery (within 1 week of the final session), and again at 12 weeks follow-up. The questionnaire will take students no more than 20-25 minutes to complete. Students will complete questionnaires under standardised conditions supervised by their teachers and trained research staff. Blinding of students, teachers, and researchers is not possible due to the nature of the intervention. However, risk of bias from teachers and researchers is minimised due to anonymous self-report assessments. Risk of contagion is also minimised by randomising at the school level. Participating schools will receive a £150 honorarium. This project has received ethical approval from the University of the West of England's Faculty Research Ethics Committee.

In order to assess the fidelity of the intervention manuals, all sessions will be audio-recorded as well as observed by a researcher and rated based on adherence to lesson plans. The interventionist and observing teachers also will be asked to complete a brief form after each lesson stating which activities were completed.

To assess intervention feasibility and acceptability, interviews will be conducted with the interventionists at the end of the programme to explore their experience of delivering the body image lessons.

In the post-intervention questionnaire, students will be asked a series of questions to assess their acceptability of the intervention. Students will indicate agreement with different statements using a 5-point Likert scale, and will be asked three open-ended questions: what they liked, what they did not like, and to list three things they learnt from the intervention.

ELIGIBILITY:
Inclusion Criteria (school):

* Co-educational secondary schools in New Delhi
* Middle income schools or private schools
* have sufficient proficiency in speaking, reading and writing in Hinglish

Exclusion Criteria (school)

* single-sex schools
* low-income schools
* do not have sufficient proficiency in speaking, reading or writing in Hinglish

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 568 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in body esteem over time: Body Esteem Scale for adolescents & adults (Mendelson, Mendelson & White, 2001). | Baseline, post-intervention (6-weeks post baseline), 10-week follow-up
  Assessment of body esteem using Body Esteem Scale for adolescents & adults,18 items, 5-point Likert-type scale. Once the appropriate items are reverse coded, scores on all items are averaged; with lower scores indicating lower body esteem.

SECONDARY OUTCOMES:
Change in eating pathology over time: Eating Disorder Examination Questionnaire (Fairburn & Beglin, 2008) | Baseline, post-intervention (6-weeks post baseline), 10-week follow-up
  Assessment of eating disorder pathology using Eating Disorder Examination Questionnaire, 28 items, 7-point Likert-type scale. Scores on all items are averaged; with higher scores indicating greater eating pathology
Internalisation of appearance ideals: The Sociocultural Attitudes Towards Appearance scale-3 (SATAQ-3): General Subscale (Thompson, Van Den Berg, Roehrig, Guarda, & Heinberg, 2004). | Baseline, post-intervention (6-weeks post baseline), 10-week follow-up
  Assessment of internalisation of appearance ideals using The Sociocultural Attitudes Towards Appearance scale-3 (SATAQ-3): General Subscale, 9 items, mean score range 1-5. Scores are averaged, with higher scores indicating higher internalisation
Life engagement Scale (Atkinson & Diedrichs, Manuscript in Preparation) | Baseline, post-intervention (6-weeks post baseline), 10-week follow-up
  Purpose-built measure assessing the extent that worries or feeling bad about the way you look has stopped you, or are likely to stop you, from engaging in life activities (e.g., going to a social event, doing physical activity, giving an opinion, going to school), 10 items, mean score range 1-4. Scores on all items are averaged; with higher scores indicating greater avoidance of activities due to appearance concerns
Positive and Negative Affect: The Positive and Negative Affect Scale (Crawford & Henry, 2004) | Baseline, post-intervention (6-weeks post baseline), 10-week follow-up
  Positive and Negative affect schedule- short form, 10 items, mean score range 1-5. Scores on the five items for the Positive Affect and Negative Affect subscales are averaged; with higher scores indicating greater negative affect and positive affect.
Self-Esteem: The Self-Esteem Scale (Rosenberg, 1965) | Baseline, post-intervention (6-weeks post baseline), 10-week follow-up
  Assessment of self-esteem using the Short-Form Rosenberg Self-Esteem scale, 10 items, mean score range 1-5. Scores are averaged, with higher scores indicating greater self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Phillippa C Diedrichs, PhD, Principal Investigator — University of the West of England
Locations (1):
- University of the West of England, Bristol, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Sabbah H, Vereecken CA, Elgar FJ, Nansel T, Aasvee K, Abdeen Z, Ojala K, Ahluwalia N, Maes L. Body weight dissatisfaction and communication with parents among adolescents in 24 countries: international cross-sectional survey. BMC Public Health. 2009 Feb 6;9:52. doi: 10.1186/1471-2458-9-52. PMID 19200369
- [Background] Fay K, Lerner RM. Weighing in on the issue: a longitudinal analysis of the influence of selected individual factors and the sports context on the developmental trajectories of eating pathology among adolescents. J Youth Adolesc. 2013 Jan;42(1):33-51. doi: 10.1007/s10964-012-9844-x. Epub 2012 Oct 31. PMID 23111843
- [Background] Wichstrom L, von Soest T. Reciprocal relations between body satisfaction and self-esteem: A large 13-year prospective study of adolescents. J Adolesc. 2016 Feb;47:16-27. doi: 10.1016/j.adolescence.2015.12.003. Epub 2015 Dec 20. PMID 26713411
- [Background] Neumark-Sztainer D, Paxton SJ, Hannan PJ, Haines J, Story M. Does body satisfaction matter? Five-year longitudinal associations between body satisfaction and health behaviors in adolescent females and males. J Adolesc Health. 2006 Aug;39(2):244-51. doi: 10.1016/j.jadohealth.2005.12.001. PMID 16857537
- [Background] Yager Z, Diedrichs PC, Ricciardelli LA, Halliwell E. What works in secondary schools? A systematic review of classroom-based body image programs. Body Image. 2013 Jun;10(3):271-81. doi: 10.1016/j.bodyim.2013.04.001. Epub 2013 May 14. PMID 23683611
- [Background] Muehlenkamp JJ, Brausch AM. Body image as a mediator of non-suicidal self-injury in adolescents. J Adolesc. 2012 Feb;35(1):1-9. doi: 10.1016/j.adolescence.2011.06.010. Epub 2011 Jul 20. PMID 21777971
- [Background] Singh MM, Ashok L, Binu VS, Parsekar SS, Bhumika TV. Adolescents and Body Image: A Cross Sectional Study. Indian J Pediatr. 2015 Dec;82(12):1107-11. doi: 10.1007/s12098-015-1768-5. Epub 2015 May 8. PMID 25947266
- [Background] Som N, Mishra SK, Mukhopadhyay S. Weight concerns and food habits of adolescent girls in two contrasting ecological regions: A comparative study in India. Eat Behav. 2016 Jan;20:21-6. doi: 10.1016/j.eatbeh.2015.11.006. Epub 2015 Nov 12. PMID 26599837
- [Background] Peltzer K, Pengpid S, James C. The globalization of whitening: prevalence of skin lighteners (or bleachers) use and its social correlates among university students in 26 countries. Int J Dermatol. 2016 Feb;55(2):165-72. doi: 10.1111/ijd.12860. Epub 2015 Oct 15. PMID 26472662
- [Background] Diedrichs PC, Atkinson MJ, Garbett KM, Leckie G. Evaluating the "Dove Confident Me" Five-Session Body Image Intervention Delivered by Teachers in Schools: A Cluster Randomized Controlled Effectiveness Trial. J Adolesc Health. 2021 Feb;68(2):331-341. doi: 10.1016/j.jadohealth.2020.10.001. Epub 2020 Nov 24. PMID 33243723
- [Background] Schrick, B. H., Sharp, E. A., Zvonkovic, A., & Reifman, A. (2012). Never let them see you sweat: Silencing and striving to appear perfect among US college women. Sex Roles, 67(11-12), 591-604.
- [Background] Ramseyer Winter, V., Kennedy, A. K., & O'Neill, E. (2017). Adolescent Tobacco and Alcohol Use: The Influence of Body Image. Journal of Child & Adolescent Substance Abuse, 26(3), 219-228.
- [Background] Dhillon, M., & Deepak, S. (2017). A body-image based media literacy intervention for Indian adolescent females. Journal of Indian Association for Child & Adolescent Mental Health, 13(1).
- See also: Girlguiding. (2016). Girls' Attitudes Survey. — http://www.girlguiding.org.uk/globalassets/docs-and-resources/research-and-campaigns/girls-attitudes-survey-2017.pdf